CLINICAL TRIAL: NCT06479668
Title: Characterize the Links Between Sleep, Emotional Dysregulation and Learning in Neurodevelopmental Disorders.
Acronym: SOM-EMO-TND
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 9094
Record Dates: First submitted 2024-06-21; First posted 2024-06-28 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-06

CONDITIONS: Attention Deficit Disorder With or Without Hyperactivity (ADHD); Autism Spectrum Disorder (ASD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autism Spectrum Disorder (Experimental)
  Interventions: Behavioral: Trier Social Stress Task
- Attention Deficit Disorder with or without Hyperactivity (Experimental)
  Interventions: Behavioral: Trier Social Stress Task

INTERVENTIONS:
Behavioral: Trier Social Stress Task — Specify details not covered in associated Arm Description.

SUMMARY:
The aim of this protocol is to disentangle the links between symptoms of emotion dysregulation, sleep disorders and cognitive deficits by measuring the effects of an emotional induction task on childrens' sleep with autism spectrum disorders (ASD) and attention deficit hyperactivity disorder (ADHD).

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 7 to 12
* Able to receive clear, age-appropriate information and to participate fully in the study
* Whose legal representative(s) are able to understand the objectives and risks of the research and to give their dated and signed informed consent.
* Subjects benefiting from a social health insurance plan (beneficiary of the legal representative(s))
* With a diagnosis made prior to inclusion of Autism Spectrum Disorder (ASD) or Attention Deficit Disorder with or without Hyperactivity (ADHD) as defined by Diagnostic and Statistical Manual 5 (DSM-5).
* With abbreviated intelligence quotient > 80 measured by Wechsler Intelligence Scale for Children version IV (WISC-IV )no more than 6 months prior to research inclusion
* No diagnosis of: fragile X syndrome, Rett syndrome, trisomy 21, tuberous sclerosis of Bourneville, von Recklinghausen disease, Cytomegalovirus encephalitis (CMV encephalitis), congenital rubella, phenylketonuria
* No clinically significant abnormality which, in the investigator's opinion, could interfere with the implementation of the study.

Exclusion Criteria:

- Current or past neurological problem(s) (e.g. stroke, epilepsy, meningitis, head trauma with loss of consciousness of more than 15 min, concussion, brain tumor, ...).

tumor, ...)

* Transmeridian travel (> 2 time zones) in the month prior to study inclusion
* Presence of a mood disorder (bipolar disorder or depression) according to DSM-5 criteria
* Social jet-lag > 2 hours (mid-point of sleep differential during weekends vs. weekdays)
* Modification of psychotropic medication in the 2 months prior to inclusion
* Use of melatonin-based dietary supplement(s)/medication(s) in the 24 hours prior to study inclusion
* Use of psychostimulant(s) within 48 hours of study entry
* Extreme chronotype (Morningness/Eveningness questionnaire score < 10 or > 42)
* Cognitive-behavioral therapies (CBT) targeting sleep disorders
* Participation in research involving an experimental drug which may interfere with the protocol*.
* Minor under guardianship
* Subject in a period of exclusion (determined by a previous or current study)
* Subject in emergency situation

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
change micro-awakening index | At Day 0 and Day 3
  polysomnography

IPD SHARING:
Plan to Share IPD: No